CLINICAL TRIAL: NCT06183567
Title: The Effect of Sedoanalgesia and General Anaesthesia on Early Neurological Recovery in Acute Ischaemic Stroke Patients Undergoing Endovascular Thrombectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, Head of Anesthesiology and Reanimation department,Assoc Prof, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UERH-AR-ZT-04
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke; Anesthesia; Neurologic Symptoms
Keywords: general anesthesia; sedoanalgesia; neurological outcome
MeSH Terms: conditions — Ischemic Stroke; Neurologic Manifestations | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Patients were divided into two groups as sedoanalgesia group (SA=31 patients) and general anesthesia group (GA=31 patients).
Who Masked: Participant, Investigator
Masking Description: The study was double-blinded, patients were selected by closed envelope method, and different clinicians administered anesthesia and postoperative follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedoanalgesia (SA) group (Active Comparator): The aim was to achieve a moderate level of sedoanalgesia (previously called conscious sedation) that would reduce agitation, anxiety and mobility but allow communication with the patient. Sedation was maintained at a level where cardiovascular function was preserved and no intervention was required to protect the airway in spontaneous breathing. Fentanyl iv 25-50 µg bolus was administered to each patient undergoing sedoanalgesia. For maintenance of sedoanalgesia, propofol iv infusion was started at doses of 1-2 mg kg-1 hour. It was titrated according to BIS level. In case of patient noncompliance, propofol iv 0.5 mg kg-1 was intervened.
  Interventions: Procedure: Sedoanalgesia; Procedure: general anesthesia
- General anesthesia (GA) group (Active Comparator): Anesthesia induction was performed with lidocaine iv 0.5 mg kg-1, propofol iv 1-2 mg kg-1, fentanyl iv 25-50 µg. After providing adequate ventilation with a mask, rocuronium iv 0.45-0.6 mg kg-1 is administered and endotracheal intubation is performed. After intubation is confirmed with end-tidal CO2 monitoring, tidal volume is set to 6-8 ml kg-1 and respiratory frequency to 12/min in CMV mode. In order to maintain cerebral perfusion, PaCO2: 35-40 mmHg is aimed to be maintained. Sevoflurane MAC 0.8 and remifentanil infusion 0.03 µg kg-1 min iv were used for maintenance of anesthesia. At the end of the procedure, sugammadex iv 2mg kg-1 was administered for extubation.
  Interventions: Procedure: Sedoanalgesia; Procedure: general anesthesia

INTERVENTIONS:
Procedure: Sedoanalgesia — In Acute Ischemic Stroke Patients Undergoing Endovascular Thrombectomy, the procedure was performed under sedoanalgesia. The procedure was continued with mean arterial pressure, heart rate, pulse oximetry and BIS monitoring.
Procedure: general anesthesia — In Acute Ischemic Stroke Patients Undergoing Endovascular Thrombectomy, the procedure was performed under general anesthesia. The procedure was continued with mean arterial pressure, heart rate, pulse oximetry and BIS monitoring.

SUMMARY:
The hypothesis of this study is that sedoanalgesia will provide better early neurological recovery than general anaesthesia in acute ischaemic stroke patients undergoing endovascular thrombectomy and to investigate the haemodynamic data of both anaesthetic methods.

DETAILED DESCRIPTION:
Endovascular mechanical thrombectomy (EMT) is the standard emergency treatment for patients presenting with acute ischemic stroke in the anterior circulation due to urgent large vessel occlusion and suitable for interventional procedures. However, despite reperfusion of the ischemia-affected area, some patients do not recover clinically. The reason for this is not known exactly. It is known that age and baseline function, which are thought to indicate brain reserve, affect the long-term outcome of stroke. Chronic hypertension, diabetes mellitus, dyslipidemia and coronary artery disease, which are associated with low brain reserve, are quite common in acute ischemic stroke patients.

There is controversy as to whether general anesthesia (GA) or sedoanalgesia (SA) should be used during EMT for acute ischemic stroke. There are not enough randomized trials addressing this question. Benefits of GA include airway preservation, pain control and potentially improved radiographic imaging and patient immobility for intervention. Conversely, GA is time-consuming and possibly associated with longer time for groin puncture and revascularization. In addition, hypotension may occur during GA, which carries a greater risk of ischemic damage. Advantages of SA may include shorter time to revascularization, fewer hemodynamic problems and the possibility of better neurological assessment during the procedure. The main arguments against SA are that patient movement can lead to procedural complications, higher radiation dose, the need for more contrast media and lack of airway control. Simonsen et al. compared general anesthesia and conscious sedation in patients with acute ischemic stroke undergoing endovascular treatment (GOLIATH) and showed that the choice of different anesthesia method can affect infarct area growth, clinical outcomes, and important physiological and anesthetic parameters.

Again, in the SIESTA (Sedation vs Intubation for Endovascular Stroke Treatment) study comparing sedation and intubation in endovascular stroke treatment, no significant difference was shown between both groups when early neurological recovery was compared (24th hour NIHSS). In this study, no superiority of conscious sedation over general anesthesia was demonstrated.

In the ESCAPE and SWIFT study, general anesthesia and conscious sedation were compared and conscious sedation was associated with better outcome than general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of cerebral ischemic embolism within the first 6 hours
2. ASA 1-4
3. Body mass index below 30 kg m-2
4. NIHSS score ≥ 10
5. Presence of isolated/combined occlusion at any level of the anterior circulation internal carotid or middle cerebral artery

Exclusion Criteria:

* Chronic renal failure
* EF less than 40
* Presence of intracranial hemorrhage
* Previous known history of severe neurological disease
* Presence of bleeding diathesis
* Pre-procedure GCS ≤ 8 and intubated patients
* Failure to clearly show the site of vascular occlusion on diagnostic imaging results
* Clinical or imaging evidence of vascular occlusion that is not internal carotid artery or middle cerebral artery
* Absence of gag reflex, loss of airway protective reflex, inadequate saliva swallowing
* History of lung infection, advanced COPD or respiratory failure
* Known history of aspiration due to vomiting,
* Known history of difficult airway
* In the presence of known intolerance or allergy to certain drugs for sedation, analgesia or both
* Previously known carotid artery stenosis
* Pregnant patients
* Patients without consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
scoring systems of neurological findings | Before Endovascular Thrombectomy and after 48 hours
  NIHSS (National Institutes of Health Stroke Scale), Glasgow coma scale (GCS) and FOUR (Full Outline of UnResponsiveness) scores
effects of both anesthesia management on hemodynamics during the procedure | Before the Endovascular Thrombectomy procedure and until the end of the recovery period (4 hours)
  Mean arterial pressure, heart rate

SECONDARY OUTCOMES:
early neurological outcome findings | 48 hours
  hemiparesis, hemiplegia, aphasia, facial paralysis
mortality and morbidity | hospitalization days
  exitus,discharge to home or palliative unit

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No